CLINICAL TRIAL: NCT05180838
Title: Remote Data Capture of Elevated Temperature Data for Early Detection of Febrile Neutropenia in Patients With Hematologic Malignancies
Brief Title: Remote Temperature Data for Early Detection of Febrile Neutropenia
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: BioIntelliSense, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-2517.cc
Record Dates: First submitted 2021-11-12; First posted 2022-01-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Hematologic Malignancy
Keywords: Cytotoxic Chemotherapy; Stem cell transplant; CAR T-cell treatments
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BioSticker: This cohort will place BioStickers at least 3 days prior to completion of standard of care therapy and discharge home post therapy.
  Interventions: Device: BioSticker

INTERVENTIONS:
Device: BioSticker — The BioSticker is an FDA approved medical device which can be worn on the upper left chest for remote data capture and can provide for up 30 days of continuous vital sign monitoring

SUMMARY:
BioSticker data is remotely tracked and displayed in a report termed the BioReport for retrospective data analysis. Typically, the biosensor collects data on an interval of ~1 minute and this data is collated and reported remotely back to the BioReport every 6 hours. More importantly, for future applications of the BioSticker for early detection of FN, there are ongoing efforts to implement real time reporting and alarms using remote monitoring services that could alert the patient that they need to seek medical care. There are no known deleterious effects from the BioSticker and it is now being widely used and tested in diverse applications including detection and contact tracing of COVID and others.

DETAILED DESCRIPTION:
The BioIntelliSense BioSticker potentially offers a solution to these challenges through early and reliable detection of elevated temperature and perhaps other relevant physiologic changes. The BioSticker is an FDA approved medical device which can be worn on the upper left chest for remote data capture and can provide for up 30 days of continuous vital sign monitoring (see https://biointellisense.com as well as attached documents on BioSticker instructions for a full description and use instructions). The BioSticker detects the following:

* Respiratory rate, heart rate at rest and skin temperature
* Body position, activity levels, sleep status
* High-resolution gait analysis and fall detection
* Symptomatic events

BioSticker data is remotely tracked and displayed in a report termed the BioReport for retrospective data analysis. Typically, the biosensor collects data on an interval of ~1 minute and this data is collated and reported remotely back to the BioReport every 6 hours. More importantly, for future applications of the BioSticker for early detection of FN, there are ongoing efforts to implement real time reporting and alarms using remote monitoring services that could alert the patient that they need to seek medical care. There are no known deleterious effects from the BioSticker and it is now being widely used and tested in diverse applications including detection and contact tracing of COVID and others.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80 years (inclusive)
* Provision to sign and date the consent form.
* Diagnosed with a hematologic malignancy and undergoing cytotoxic chemotherapy, stem cell transplants or CAR T-cell treatments at the Blood Disorders and Cell Therapies Center at UCHealth (BDCTC)
* Will have longitudinal care provided by the BDCTC for >1 additional month
* Receive chemotherapy or other therapies known to cause reductions in WBC <1000 on a routine basis
* Scheduled to be discharged home and self-monitor for FN and other complications
* Patient is willing to tell TSA or any security representative that you are wearing a "medical device"
* Patient has agreed to not submerge the device underwater including while swimming or bathing
* Patient is willing to complete a self-check temperature log comply and be available for the duration of the study
* Patient has access to a thermometer

Exclusion Criteria:

* Patient that wears a defibrillator, pacemaker, or other implantable device
* Patient has broken skin including wounds, sores, or abrasions in the area that the BioSticker would be applied
* Patient has had a severe reaction to silicone adhesives
* Patient has any clinically significant medical or psychiatric disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with leukemia, lymphoma, myeloma and other blood cancers undergoing treatment with cytotoxic chemotherapy, stem cell transplant or CAR T-cells following IRB consent. Patients will be included who are >18 years old, will have longitudinal care provided by the BDCTC for >1 additional month, receive chemotherapy or other therapies known to cause reductions in WBC <1000 on a routine basis, are capable of informed consent and agree to collect a self-check temperature log.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Reliability of BioSticker compared to self-check | 28 days
  Patients will self-temperature check every 6 hours or at least two times per day, and will log these temperatures in a paper record with date, time and temperature noted.

SECONDARY OUTCOMES:
BioSticker Impact on Patient reported temperature | 28 days
  Patients will report a single oral temperature of ≥38.3°C (101°F) or a temperature of ≥38.0°C (100.4°F) sustained over a one-hour period to our clinic nurses or 24/7 on-call advanced practitioner and will be directed to the Emergency Department or clinic for initiation of antibiotics and FN work-up and management as per usual practice.
BioSticker Impact on Length of Hospitalization | 28 days
  Hospitalization during the 28 days will be extracted from the medical record
BioSticker Impact on ICU transfers | 28 days
  ICU transfers during the 28 days will be extracted from the medical record
BioSticker Impact on Delays in Chemotherapy | 28 days
  Delays in chemotherapy during the 28 days will be extracted from the medical record

CONTACTS AND LOCATIONS:
Overall Officials: Glen Peterson, Principal Investigator — Colorado Research Center
Locations (2):
- United States (2):
  - Colorado Research Center, Aurora, Colorado
  - UCHealth-Metro Denver, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No